CLINICAL TRIAL: NCT07017244
Title: Randomized Double-blind Monocentric Clinical Trial on the Effect of a Dietary Supplement vs Low-dosage Product on Reduction of Infant Gastrointestinal Discomfort and Colics
Brief Title: Effect of a Dietary Supplement vs Low-dosage Product on Infant Gastrointestinal Discomfort and Colics
Acronym: DISIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENTEROBABY
Record Dates: First submitted 2025-05-06; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Infant Colic; Gut Microbiota
MeSH Terms: conditions — Colic | interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Intervention Model Description: Prospective Randomized and Double-Blind Controlled Vs Low-dosage product
Who Masked: Participant, Care Provider
Masking Description: Different batch code assigned to products, same labeling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): Partecipants received Enterobaby, a food supplement based on a mixture of Lactobacillus acidophilus DSM 25175, Lactobacillus reuteri DSM 24936, Matricaria chamomilla L. oleolite, extra-virgin olive oil in oral suspension
  Interventions: Dietary Supplement: Verum
- Low-dosage product (Active Comparator): Partecipants received a food supplement based on a mixture of maltodextrine, Magnesium stearate and Sun flower oil and less than 0,1% of Lactobacillus acidophilus DSM 25175 and Lactobacillus reuteri DSM 24936, 1% of Matricaria chamomilla L. oleolite and extra-virgin olive oil in oral suspension
  Interventions: Dietary Supplement: Active comparator

INTERVENTIONS:
Dietary Supplement: Verum — 1st cycle - 30 days continuous use Cycle 2 - 30-day washout
  Arms: Verum
Dietary Supplement: Active comparator — 1st cycle - 30 days continuous use Cycle 2 - 30-day washout
  Arms: Low-dosage product

SUMMARY:
The goal of this clinical trial is to verify whether a food supplement is effective in treating infantile colic of infants aged between 21 days and 9 months and the colonization ability of the gut microbiota by measuring faecal relative abundance of the gut microbiota probiotic treatment species.

The main outcomes are: - the mean number of crying episodes and the sleep duration - Relative abundance of the gut microbiota probiotic treatment species.

DETAILED DESCRIPTION:
Infant colic, characterized by excessive crying/fussing for no apparent cause, is common and distressing to families.

The exact causes of infant colic are heterogeneous and not fully understood in detail, but some likely hypotheses point on factors such as gut dysmotility and food intolerance. Growing evidence suggests that the gut microbiota could be also involved in colics: a higher amount of Coliforms and a lower amount of Lactobacilli have been found in colicky infants compared to non-colicky subjects, and probiotic supplementation with Lactobacillus reuteri has been shown to be effective in treating the condition in some clinical trials of breastfed infants.

In the present study, the investigator performs a randomized controlled clinical trial aimed to verify whether a food supplement is effective in treating infantile colic of infants and colonization ability of the gut microbiota by measuring faecal relative abundance of the gut microbiota probiotic treatment species.

The product is a food supplement based on freeze-dried probiotics (Lactobacillus reuteri DSM 25175 and Lactobacillus acidophilus DSM 24936) and chamomile oleolite to promote the balance of the intestinal bacterial flora, on gastrointestinal discomfort in children aging 0-9 months.

Treatment consists of taking the product or the low-dosage product 7 drops x 2/die for a 30-days. A follow-up was made after 30 days wash out.

Infant colics are diagnosed with FLACC (Face, Legs, Activity, Cry, Consolability

* preverbal patient pain scale) and G4 Infant Colic Rome IV criteria, while relative abundance of the gut microbiota probiotic treatment species (L. reuteri and L. acidophilus) will be evaluated using quantitative PCR (Polymerase Chain Reaction), in order to identify the colonization ability of the study treatment (Fecal sample).

ELIGIBILITY:
Inclusion Criteria:

* Children Age: 0-9 months Infant colics diagnosed with FLACC (Face, Legs, Activity, Cry, Consolability - preverbal patient pain scale) and G4 Infant Colic Rome IV criteria

Exclusion Criteria:

* infants suffering from acute or chronic diseases, such as chronic lung disease; diarrhea underlying specific diseases or developmental disorders confirmed by a pediatrician
* infants participating in other clinical studies
* age ≥ 9 months
* neurological diseases
* suspected or confirmed food allergy to the ingredients of the products under study
* gastroesophageal reflux disease
* use of antibiotics 1-2 weeks before enrolment
* use of gastric acidity inhibitors at any time before enrolment
* fever and/or infectious diseases at any time before enrolment
* current systemic infections
* history of congenital infections

Ages: 0 Months to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of infant gastrointestinal discomfort and colics by measuring the medium full-force daily crying | T0 (first visit) - T1 (after 7 days) - T2 (after 15 days) - T3 (after 30 days) - T4 (after 60 days)
  The mean daily minutes of crying will be calculated as a sum of crying, fussing, and unsuitable crying using a parental diary.

SECONDARY OUTCOMES:
Evaluation of relative abundance of the gut microbiota probiotic treatment species | Faecal samples will be collected from each subject before starting supplementation, at the end of the study period T3 (30 days) and at T4 (after 30 days wash out) and will be analyzed.
  Relative abundance of the gut microbiota probiotic treatment species (L. reuteri and L. acidophilus) will be evaluated using quantitative PCR (Polymerase Chain Reaction), in order to identify the colonization ability of the study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Gioacchino Calapai, Messina, Italy